CLINICAL TRIAL: NCT03921424
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by Administration of PNEUMOVAX™23 Eight Weeks Later in Children Infected With Human Immunodeficiency Virus (HIV) (PNEU-WAY PED)
Brief Title: Safety and Immunogenicity of V114 in Children Infected With Human Immunodeficiency Virus (HIV) (V114-030/PNEU-WAY PED)
Acronym: PNEU-WAY PED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V114-030; V114-030 (Other: Merck); 2019-000341-12 (EudraCT Number)
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal conjugate vaccine (PCV), 15-valent, 22F, 33F
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2)
  Interventions: Biological: V114; Biological: PNEUMOVAX™23
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2)
  Interventions: Biological: Prevnar 13™; Biological: PNEUMOVAX™23

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) present in Prevnar 13™ plus 2 additional serotypes (22F, 33F) in each 0.5 mL dose.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Biological: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) in each 0.5 mL dose.
  Arms: Prevnar 13™
Biological: PNEUMOVAX™23 — 23-valent pneumococcal polysaccharide vaccine containing 23 serotypes (1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F) in each 0.5 mL dose

SUMMARY:
This is a study of V114 in children infected with HIV. Participants will be randomly assigned in a 1:1 ratio to receive either V114 or Prevnar 13™ followed 8 weeks later by a single dose of PNEUMOVAX™23. The primary objectives of this study are to evaluate the safety and tolerability of V114 in children 6 to 17 years of age inclusive infected with HIV and to evaluate the anti-pneumococcal polysaccharide (PnPs) serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) at 30 days following vaccination with V114 or Prevnar 13™ by each vaccination group. There are no formal hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 6 and 17 years (inclusive) infected with HIV and has a Cluster of Differentiation 4+ (CD4+) T-cell count ≥200 cells/µL and plasma HIV ribonucleic acid (RNA) <50,000 copies/mL
* Is Pneumococcal Conjugate Vaccine (PCV) naïve, previously vaccinated with a <13-valent PCV, partially vaccinated with Prevnar 13™, or has a history of previous Prevnar 13™ vaccination ≥3 years before Visit 2 (Day 1)
* Is PnPs vaccine naïve or has a history of 1 previous PnPs vaccination ≥5 years before Visit 2 (Day 1)
* Female participant: not pregnant, not breastfeeding and 1) not of childbearing potential, or 2) of childbearing potential and agrees to practice contraception through 6 weeks after administration of last dose of the study vaccine.

Exclusion Criteria:

* History of World Health Organization (WHO) HIV classification of clinical Stage 4 disease within the past 12 months
* History of invasive pneumococcal disease
* Known hypersensitivity to any vaccine component
* Known or suspected congenital immunodeficiency (other than HIV infection), functional or anatomic asplenia, or history of autoimmune disease
* Bleeding disorder contraindicating intramuscular vaccinations
* History of malignancy ≤5 years prior to signing informed consent/assent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Female participant: positive urine or serum pregnancy test
* Expect to receive any pneumococcal vaccine during the study outside of the protocol
* Receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received a blood transfusion or blood products within 6 months of enrollment
* Participated in another clinical study of an investigational product within 2 months of enrollment
* Current user of recreational or illicit drugs or history of drug or alcohol abuse or dependence

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 407 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- South Africa (4):
  - Perinatal HIV Research Unit ( Site 0042), Johannesburg, Gauteng
  - Wits Reproductive Health and HIV Institute (WRHI) ( Site 0043), Johannesburg, Gauteng
  - Family Clinic Research With UBUNTU ( Site 0045), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 0041), Paarl, Western Cape
- Thailand (4):
  - Chulalongkorn University-Pediatrics ( Site 0062), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Pediatric Infectious Diseases ( Site 0064), Bangkok, Bangkok
  - Faculty of Medicine - Khon Kaen University-Pediatrics ( Site 0063), Amphoe Mueang, Changwat Khon Kaen
  - CM Clinical Trial Unit-CM Clinical Trial Unit ( Site 0061), Chiang Mai
- Ukraine (5):
  - Community Instit Dnipropetrovsk Municipal clinical Hospital #21 ( Site 0088), Dnipro, Dnipropetrovsk Oblast
  - Dnipropetrovsk Regional Center of Socially Significant Diseases ( Site 0082), Dnipro, Dnipropetrovsk Oblast
  - Odesa Regional Center of Socially Significant Diseases ( Site 0083), Odesa, Odesa Oblast
  - Vinnitsa Reg Cntr for AIDS Prevention-Control-Outpatient clinic dept ( Site 0086), Vinnytsia, Vinnytsia Oblast
  - Zaporizhzhya Regional Clinical Children's Hospital ( Site 0089), Zaporizhzhya, Zaporizhzhia Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wilck M, Barnabas S, Chokephaibulkit K, Violari A, Kosalaraksa P, Yesypenko S, Chukhalova I, Dagan R, Richmond P, Mikviman E, Morgan L, Feemster K, Lupinacci R, Chiarappa J, Madhi SA, Bickham K, Musey L; V114-030 Study Group. A phase 3 study of safety and immunogenicity of V114, a 15-valent pneumococcal conjugate vaccine, followed by 23-valent pneumococcal polysaccharide vaccine, in children with HIV. AIDS. 2023 Jul 1;37(8):1227-1237. doi: 10.1097/QAD.0000000000003551. Epub 2023 Mar 17. PMID 36939067

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 407 participants were randomized in a 1:1 ratio to receive either V114 or Prevnar 13™ on Day 1 and PNEUMOVAX™23 at Week 8.
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2).
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 203 | 204
Vaccination 1 - (Day 1) | 203 | 204
Vaccination 2 - (Week 8) | 203 | 202 (Two participants did not receive Vaccination 2.)
Completed | 203 | 201
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal By Parent/Guardian | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 203 | 204 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.7) | 12.6 (3.0) | 12.7 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 60 | 62 | 122
  Adolescents (12-17 years) | 143 | 142 | 285
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 99 | 195
  Male | 107 | 105 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 201 | 203 | 404
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 66 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 88 | 78 | 166
  White | 40 | 49 | 89
  More than one race | 12 | 9 | 21
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-Site Adverse Event Following Vaccination With V114 or Prevnar 13™
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following Vaccination 1 with either V114 or Prevnar 13™, the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were redness/erythema, hard lump/induration, tenderness/pain, and swelling.
Time Frame: Through 14 Days after Vaccination 1 (Up to Day 14)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 204
Percentage of Participants
  Injection site redness/erythema | 9.4 (5.7) [5.7 to 14.2] | 5.9 (3.1) [3.1 to 10.0]
  Injection site hard lump/induration | 10.3 (6.5) [6.5 to 15.4] | 6.4 (3.4) [3.4 to 10.7]
  Injection site tenderness/pain | 55.2 (48.1) [48.1 to 62.1] | 53.9 (46.8) [46.8 to 60.9]
  Injection site swelling | 28.6 (22.5) [22.5 to 35.3] | 21.6 (16.1) [16.1 to 27.9]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event Following Vaccination With V114 or Prevnar 13™
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following Vaccination 1 with either V114 or Prevnar 13™, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were joint pain/arthralgia, tiredness/fatigue, headache, muscle pain/myalgia, and hives or welts/urticaria.
Time Frame: Through 14 Days after Vaccination 1 (Up to Day 14)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 204
Percentage of Participants
  Joint pain/arthralgia | 9.4 (5.7) [5.7 to 14.2] | 10.3 (6.5) [6.5 to 15.3]
  Tiredness/fatigue | 7.9 (4.6) [4.6 to 12.5] | 8.3 (4.9) [4.9 to 13.0]
  Headache | 14.8 (10.2) [10.2 to 20.4] | 10.8 (6.9) [6.9 to 15.9]
  Muscle pain/myalgia | 34.0 (27.5) [27.5 to 41.0] | 25.5 (19.7) [19.7 to 32.0]
  Hives or welts/urticaria | 0.5 (0.0) [0.0 to 2.7] | 1.5 (0.3) [0.3 to 4.2]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event (SAE) Following Vaccination 1 (V114 or Prevnar 13™) or Vaccination 2 (PNEUMOVAX™23) Through Completion of Study
Description: An SAE is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is an other important medical event deemed such by medical or scientific judgment. The percentage of participants with a vaccine-related SAE following Vaccination 1 (with either V114 or Prevnar 13™) or Vaccination 2 (PNEUMOVAX™23) through completion of study participation was reported.
Time Frame: Through 6 Months after Vaccination 1 (Up to Day 194)
Population: All randomized participants who received at least 1 dose of the relevant study vaccination for the timepoint of interest were analyzed. Two participants in the Prevnar 13™ group did not receive PNEUMOVAX™23 and therefore were not analyzed for Vaccination 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 204
Percentage of Participants
  Vaccination 1 | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 1.8]
  Vaccination 2: number analyzed (Participants) | 203 | 202
  Vaccination 2 | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 1.8]

4. Primary Outcome: Anti-PnPs Serotype-specific IgG Geometric Mean Concentrations (GMCs) at 30 Days Following Vaccination With V114 or Prevnar 13™
Description: The GMC of serotype-specific IgG for the serotypes contained in V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay.
Time Frame: Day 30
Population: All randomized participants included participants without protocol deviations that could have substantially impacted the results of the immunogenicity outcome measure and who had sufficient serum volume to perform the analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 204
μg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 194 | 196
  Serotype 1 (Shared) | 2.17 [1.89 to 2.48] | 3.26 [2.82 to 3.77]
  Serotype 3 (Shared): number analyzed (Participants) | 194 | 196
  Serotype 3 (Shared) | 1.05 [0.93 to 1.19] | 0.84 [0.73 to 0.97]
  Serotype 4 (Shared): number analyzed (Participants) | 194 | 196
  Serotype 4 (Shared) | 2.59 [2.23 to 3.00] | 4.27 [3.57 to 5.11]
  Serotype 5 (Shared): number analyzed (Participants) | 194 | 196
  Serotype 5 (Shared) | 2.94 [2.44 to 3.54] | 2.78 [2.30 to 3.37]
  Serotype 6A (Shared): number analyzed (Participants) | 194 | 196
  Serotype 6A (Shared) | 7.98 [6.30 to 10.11] | 7.56 [6.06 to 9.45]
  Serotype 6B (Shared): number analyzed (Participants) | 194 | 196
  Serotype 6B (Shared) | 11.44 [9.07 to 14.43] | 6.92 [5.45 to 8.79]
  Serotype 7F (Shared): number analyzed (Participants) | 194 | 196
  Serotype 7F (Shared) | 4.84 [4.10 to 5.71] | 5.00 [4.29 to 5.83]
  Serotype 9V (Shared): number analyzed (Participants) | 194 | 196
  Serotype 9V (Shared) | 4.15 [3.56 to 4.85] | 4.78 [4.03 to 5.66]
  Serotype 14 (Shared): number analyzed (Participants) | 194 | 196
  Serotype 14 (Shared) | 20.38 [16.39 to 25.35] | 18.29 [14.43 to 23.17]
  Serotype 18C (Shared): number analyzed (Participants) | 194 | 196
  Serotype 18C (Shared) | 5.18 [4.32 to 6.20] | 5.15 [4.29 to 6.18]
  Serotype 19A (Shared): number analyzed (Participants) | 194 | 196
  Serotype 19A (Shared) | 14.20 [11.81 to 17.07] | 14.78 [12.45 to 17.54]
  Serotype 19F (Shared): number analyzed (Participants) | 194 | 196
  Serotype 19F (Shared) | 9.76 [8.03 to 11.85] | 8.61 [7.28 to 10.18]
  Serotype 23F (Shared): number analyzed (Participants) | 194 | 196
  Serotype 23F (Shared) | 6.71 [5.42 to 8.31] | 6.35 [5.14 to 7.85]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 194 | 193
  Serotype 22F (Unique to V114) | 9.28 [7.76 to 11.09] | 0.24 [0.20 to 0.29]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 194 | 196
  Serotype 33F (Unique to V114) | 4.53 [3.80 to 5.39] | 0.29 [0.25 to 0.33]

5. Secondary Outcome: Percentage of Participants With a Solicited Injection-Site Adverse Event Following Vaccination With PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following Vaccination 2 with PNEUMOVAX™23 (PPV23), the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were redness/erythema, hard lump/induration, tenderness/pain, and swelling.
Time Frame: Through 14 Days after Vaccination 2 (Up to Day 84)
Population: All randomized participants who received at least 1 dose of the relevant study vaccination for the timepoint of interest were analyzed. Two participants in the Prevnar 13™ group did not receive PNEUMOVAX™23 and therefore were not included in the analysis for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 202
Percentage of Participants
  Injection site redness/erythema | 10.3 (6.5) [6.5 to 15.4] | 12.4 (8.2) [8.2 to 17.7]
  Injection site hard lump/induration | 18.2 (13.2) [13.2 to 24.2] | 13.4 (9.0) [9.0 to 18.8]
  Injection site tenderness/pain | 51.7 (44.6) [44.6 to 58.8] | 55.0 (47.8) [47.8 to 61.9]
  Injection site swelling | 47.3 (40.3) [40.3 to 54.4] | 34.7 (28.1) [28.1 to 41.7]

6. Secondary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event Following Vaccination With PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following Vaccination 2 with PNEUMOVAX™23, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were joint pain/arthralgia, tiredness/fatigue, headache, muscle pain/myalgia, and hives or welts/urticaria.
Time Frame: Through 14 Days after Vaccination 2 (Up to Day 84)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 202
Percentage of Participants
  Joint pain/arthralgia | 12.8 (8.5) [8.5 to 18.2] | 8.4 (5.0) [5.0 to 13.1]
  Tiredness/fatigue | 12.3 (8.1) [8.1 to 17.6] | 11.4 (7.4) [7.4 to 16.6]
  Headache | 10.3 (6.5) [6.5 to 15.4] | 9.4 (5.8) [5.8 to 14.3]
  Muscle pain/myalgia | 43.3 (36.4) [36.4 to 50.5] | 39.1 (32.3) [32.3 to 46.2]
  Hives or welts/urticaria | 0.0 (0.0) [0.0 to 1.8] | 0.5 (0.0) [0.0 to 2.7]

7. Secondary Outcome: Anti-PnPs Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at 30 Days Following Vaccination With V114 or Prevnar 13™
Description: The GMT of serotype-specific OPA for the serotypes contained in V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a multiplexed opsonophagocytic assay.
Time Frame: Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 204
Titers (1/dil)
  Serotype 1 (Shared): number analyzed (Participants) | 164 | 160
  Serotype 1 (Shared) | 353.4 [278.4 to 448.7] | 398.3 [313.5 to 506.1]
  Serotype 3 (Shared): number analyzed (Participants) | 163 | 158
  Serotype 3 (Shared) | 330.0 [284.4 to 383.0] | 301.5 [255.5 to 355.7]
  Serotype 4 (Shared): number analyzed (Participants) | 164 | 159
  Serotype 4 (Shared) | 6078.3 [5106.1 to 7235.4] | 9172.8 [7582.8 to 11096.1]
  Serotype 5 (Shared): number analyzed (Participants) | 164 | 160
  Serotype 5 (Shared) | 847.6 [671.1 to 1070.4] | 642.1 [490.9 to 839.9]
  Serotype 6A (Shared): number analyzed (Participants) | 163 | 159
  Serotype 6A (Shared) | 14274.6 [12014.1 to 16960.4] | 11915.4 [10160.9 to 13973.0]
  Serotype 6B (Shared): number analyzed (Participants) | 164 | 160
  Serotype 6B (Shared) | 17636.5 [14728.7 to 21118.3] | 15052.9 [12719.6 to 17814.2]
  Serotype 7F (Shared): number analyzed (Participants) | 164 | 160
  Serotype 7F (Shared) | 17574.4 [15234.2 to 20274.0] | 18519.3 [16010.9 to 21420.8]
  Serotype 9V (Shared): number analyzed (Participants) | 164 | 160
  Serotype 9V (Shared) | 4800.0 [4201.0 to 5484.4] | 5879.7 [4853.9 to 7122.2]
  Serotype 14 (Shared): number analyzed (Participants) | 164 | 160
  Serotype 14 (Shared) | 18444.3 [15257.3 to 22297.0] | 17920.8 [14874.4 to 21591.2]
  Serotype 18C (Shared): number analyzed (Participants) | 163 | 160
  Serotype 18C (Shared) | 4556.2 [3794.1 to 5471.5] | 3543.0 [2919.6 to 4299.5]
  Serotype 19A (Shared): number analyzed (Participants) | 164 | 160
  Serotype 19A (Shared) | 8176.4 [6778.3 to 9862.8] | 8690.2 [7382.3 to 10229.8]
  Serotype 19F (Shared): number analyzed (Participants) | 164 | 159
  Serotype 19F (Shared) | 3711.8 [3178.0 to 4335.2] | 3277.6 [2833.1 to 3791.8]
  Serotype 23F (Shared): number analyzed (Participants) | 162 | 160
  Serotype 23F (Shared) | 11693.1 [9483.8 to 14417.1] | 11933.8 [9597.5 to 14838.8]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 164 | 142
  Serotype 22F (Unique to V114) | 10791.3 [9157.2 to 12716.9] | 503.1 [330.1 to 766.8]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 162 | 159
  Serotype 33F (Unique to V114) | 36357.0 [31146.2 to 42439.6] | 5520.6 [4659.5 to 6540.9]

8. Secondary Outcome: Anti-PnPs Serotype-specific OPA GMTs at 30 Days Following Vaccination With PNEUMOVAX™23 (Week 12)
Description: as for outcome 7
Time Frame: Week 12
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 202
Titers (1/dil)
  Serotype 1 (Shared): number analyzed (Participants) | 164 | 162
  Serotype 1 (Shared) | 326.4 [267.0 to 399.0] | 337.0 [272.3 to 417.1]
  Serotype 3 (Shared): number analyzed (Participants) | 164 | 161
  Serotype 3 (Shared) | 327.2 [278.9 to 383.9] | 384.8 [333.0 to 444.6]
  Serotype 4 (Shared): number analyzed (Participants) | 164 | 162
  Serotype 4 (Shared) | 5445.7 [4663.7 to 6358.8] | 7526.8 [6309.7 to 8978.7]
  Serotype 5 (Shared): number analyzed (Participants) | 165 | 162
  Serotype 5 (Shared) | 985.6 [813.6 to 1193.8] | 939.5 [737.3 to 1197.3]
  Serotype 6A (Shared): number analyzed (Participants) | 164 | 162
  Serotype 6A (Shared) | 10208.7 [8703.8 to 11973.7] | 10699.8 [9010.5 to 12705.7]
  Serotype 6B (Shared): number analyzed (Participants) | 164 | 162
  Serotype 6B (Shared) | 13774.8 [11661.6 to 16271.0] | 12745.8 [10887.3 to 14921.6]
  Serotype 7F (Shared): number analyzed (Participants) | 165 | 162
  Serotype 7F (Shared) | 17415.9 [15091.4 to 20098.5] | 19140.5 [16778.5 to 21835.0]
  Serotype 9V (Shared): number analyzed (Participants) | 165 | 161
  Serotype 9V (Shared) | 5135.9 [4328.2 to 6094.3] | 6152.2 [5219.6 to 7251.4]
  Serotype 14 (Shared): number analyzed (Participants) | 165 | 161
  Serotype 14 (Shared) | 17207.5 [14074.5 to 21037.9] | 16461.2 [13695.1 to 19785.9]
  Serotype 18C (Shared): number analyzed (Participants) | 165 | 161
  Serotype 18C (Shared) | 3635.1 [3103.0 to 4258.5] | 3369.0 [2844.0 to 3990.9]
  Serotype 19A (Shared): number analyzed (Participants) | 164 | 162
  Serotype 19A (Shared) | 7613.7 [6414.6 to 9036.9] | 8838.0 [7592.6 to 10287.6]
  Serotype 19F (Shared): number analyzed (Participants) | 165 | 162
  Serotype 19F (Shared) | 3694.8 [3212.9 to 4248.9] | 3904.4 [3382.3 to 4507.1]
  Serotype 23F (Shared): number analyzed (Participants) | 163 | 161
  Serotype 23F (Shared) | 10216.7 [8465.7 to 12329.8] | 10086.0 [8334.0 to 12206.2]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 165 | 162
  Serotype 22F (Unique to V114) | 8756.1 [7419.0 to 10334.1] | 6958.0 [5941.5 to 8148.5]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 163 | 162
  Serotype 33F (Unique to V114) | 34173.6 [29554.9 to 39514.0] | 30651.0 [26240.5 to 35802.8]

9. Secondary Outcome: Anti-PnPs Serotype-specific IgG GMCs at 30 Days Following Vaccination With PNEUMOVAX™23 (Week 12)
Description: as for outcome 4
Time Frame: Week 12
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 203 | 202
μg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 192 | 183
  Serotype 1 (Shared) | 2.58 [2.31 to 2.88] | 3.33 [2.95 to 3.75]
  Serotype 3 (Shared): number analyzed (Participants) | 192 | 183
  Serotype 3 (Shared) | 1.10 [0.97 to 1.24] | 1.08 [0.94 to 1.24]
  Serotype 4 (Shared): number analyzed (Participants) | 192 | 182
  Serotype 4 (Shared) | 2.36 [2.08 to 2.69] | 3.61 [3.09 to 4.23]
  Serotype 5 (Shared): number analyzed (Participants) | 192 | 183
  Serotype 5 (Shared) | 3.01 [2.58 to 3.52] | 3.24 [2.75 to 3.82]
  Serotype 6A (Shared): number analyzed (Participants) | 192 | 183
  Serotype 6A (Shared) | 4.67 [3.74 to 5.84] | 4.91 [3.94 to 6.11]
  Serotype 6B (Shared): number analyzed (Participants) | 192 | 183
  Serotype 6B (Shared) | 7.12 [5.75 to 8.81] | 4.96 [3.96 to 6.22]
  Serotype 7F (Shared): number analyzed (Participants) | 192 | 183
  Serotype 7F (Shared) | 4.10 [3.55 to 4.72] | 4.27 [3.71 to 4.92]
  Serotype 9V (Shared): number analyzed (Participants) | 192 | 183
  Serotype 9V (Shared) | 3.69 [3.20 to 4.25] | 4.52 [3.89 to 5.24]
  Serotype 14 (Shared): number analyzed (Participants) | 192 | 183
  Serotype 14 (Shared) | 18.88 [15.43 to 23.09] | 19.89 [16.00 to 24.72]
  Serotype 18C (Shared): number analyzed (Participants) | 192 | 183
  Serotype 18C (Shared) | 3.75 [3.18 to 4.43] | 4.11 [3.48 to 4.85]
  Serotype 19A (Shared): number analyzed (Participants) | 192 | 183
  Serotype 19A (Shared) | 11.23 [9.48 to 13.31] | 12.19 [10.38 to 14.32]
  Serotype 19F (Shared): number analyzed (Participants) | 192 | 183
  Serotype 19F (Shared) | 8.56 [7.26 to 10.08] | 7.98 [6.83 to 9.33]
  Serotype 23F (Shared): number analyzed (Participants) | 192 | 183
  Serotype 23F (Shared) | 4.40 [3.63 to 5.34] | 4.83 [3.96 to 5.88]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 192 | 183
  Serotype 22F (Unique to V114) | 8.18 [7.10 to 9.42] | 10.32 [8.67 to 12.29]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 192 | 183
  Serotype 33F (Unique to V114) | 3.76 [3.23 to 4.38] | 6.18 [5.23 to 7.30]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: Up to 14 days after each vaccination; Serious adverse events and All-Cause Mortality: Through 6 months after Vaccination 1 (Up to Day 194).
Description: The analysis population for All-Cause Mortality included all randomized participants. The analysis population for AEs included all randomized participants who received at least 1 dose of study vaccination. All randomized participants received treatment. Two participants in the Prevnar 13™ group did not receive PNEUMOVAX™23.
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1).
- V114 (Post-PNEUMOVAX™23): Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2).
- Prevnar 13™ (Post-PNEUMOVAX™23): Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and were to receive a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™ | V114 (Post-PNEUMOVAX™23) | Prevnar 13™ (Post-PNEUMOVAX™23)
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/204 | 0/203 | 0/202
Serious Adverse Events (participants affected / at risk) | 1/203 | 1/204 | 2/203 | 2/202
Other Adverse Events (participants affected / at risk) | 158/203 | 138/204 | 152/203 | 154/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=203) | Prevnar 13™ (N=204) | V114 (Post-PNEUMOVAX™23) (N=203) | Prevnar 13™ (Post-PNEUMOVAX™23) (N=202)
Serous retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=203) | Prevnar 13™ (N=204) | V114 (Post-PNEUMOVAX™23) (N=203) | Prevnar 13™ (Post-PNEUMOVAX™23) (N=202)
Fatigue (General disorders) | 16 (16) | 17 (19) | 25 (30) | 23 (23)
Injection site erythema (General disorders) | 19 (20) | 12 (13) | 21 (21) | 25 (25)
Injection site induration (General disorders) | 21 (22) | 13 (13) | 37 (37) | 27 (27)
Injection site pain (General disorders) | 112 (122) | 110 (117) | 105 (110) | 111 (117)
Injection site swelling (General disorders) | 58 (59) | 44 (49) | 96 (97) | 70 (70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 21 (24) | 26 (26) | 17 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 69 (72) | 52 (56) | 88 (91) | 79 (80)
Headache (Nervous system disorders) | 30 (34) | 22 (28) | 21 (25) | 19 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03921424/Prot_SAP_000.pdf